CLINICAL TRIAL: NCT05962866
Title: Pregnancy of I. and II. Leopold Manoeuvres Performed by Pregnant Women Under Midwife Supervision Effects on Distress and Perception of Motherhood Role
Brief Title: The Effect of Pregnant Women's Maneuvers on Pregnancy Distress and Perception of Maternity Role"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel ÖZTÜRK (Other)
Responsible Party: Sponsor-Investigator, Sibel ÖZTÜRK, Asst. Prof., Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ataturk University SOZTURK0003
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy Related; Mother-Child Relations
Keywords: Leopold maneuver; pregnancy; midwifery; fetus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment: Have pregnant women perform the 1st and 2nd Leopold Maneuvers (Experimental): Voluntary information form will be read to those who want to participate in the research, verbal and written permissions will be obtained and information will be given about fetal development and Leopold maneuvers in the pregnant follow-up room of the family health center. This transaction is 28-32. 32-38 at the next follow-up at gestational weeks. Pregnancy will be carried out with the same procedure.
  Interventions: Other: I and II. Performing Leopold Maneuvers by the pregnant
- Control: Assigned Interventions standard care group (No Intervention): No intervention will be made.

INTERVENTIONS:
Other: I and II. Performing Leopold Maneuvers by the pregnant — 24-32 and 32-38 days of pregnancy by the pregnant woman. 1st and 2nd leoppold maneuvers are performed by the pregnant woman, 2 times between weeks.
  Arms: Experiment: Have pregnant women perform the 1st and 2nd Leopold Maneuvers

SUMMARY:
The role of motherhood; Motherhood can be defined as a learning process that includes knowledge, skills, attitudes and behaviors of a woman who has been handed down from generation to generation. Mother-infant attachment; At the behavioral and emotional level, it is the mother's attachment to her baby, which becomes stronger as the pregnant woman's body changes, her uterus expands and the mother begins to feel fetal movements. The fact that women adopt the role of motherhood throughout pregnancy is very important for attachment behaviors and infant attachment patterns in the early and late postpartum period.

DETAILED DESCRIPTION:
It is very important for midwives to implement and teach the interventions that will enable pregnant women to take an active role in this period, in terms of perception of the role of motherhood and pregnancy distress. . The literature provides a data source for leopard maneuvers. However, I and II. There is no study on the effect of Leopold maneuvers on pregnancy distress and the perception of maternal role. This study, which is planned to support and develop awareness in this area, is important in terms of literature.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous single pregnancy,
* 28th gestational week,
* Over the age of 18, under the age of 40,
* Not having communication difficulties and mental disabilities, Literate,
* Not having any chronic health problems (hypertension, heart disease,
* obesity etc.)
* Does not have a psychiatric disease and does not use psychiatric drugs, Exclusion Criteria
* Not open to communication and cooperation during the working period,
* Reluctant to participate in the research,
* Not completing the questionnaires,
* Pregnant women who gave birth prematurely were not included in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — being pregnant
Enrollment: 120 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Measuring pregnancy distress of pregnant women | two months
  The Cronbach Alpha value of the scale was found to be 0.83. The scale, which can be applied to pregnant women who are twelve weeks and older, consists of 16 items and is graded as a 4-point Likert scale. The total score that can be obtained from the scale ranges from 0 to 48. A total score of 28 and above according to the cut-off point indicates that the pregnant woman is at risk for distress. The scale has 2 sub-dimensions as "negative affect" consisting of 11 items and "partner participation" consisting of 5 items. Items 1, 2, 4, 8 and 15 in the scale belong to peer involvement, other items belong to negative affect.

SECONDARY OUTCOMES:
Measuring pregnant women's perception of maternal role | two months
  The internal consistency reliability of the scale was found to be between 0.81-0.85. The validity and reliability study of the scale was adapted to Turkish society by Çalışır The scale consists of 11 semantic opposite adjective pairs with 22 items and seven points, which analyze the concept of Me as a Mother. These 11 items are distributed within the 22 item opposite adjective pairs in the scale. Three items were evaluated with reverse scoring to avoid the possibility of bias while the participant was answering the questions. Items 3, 7 and 8 were evaluated over 1 point instead of 7 points. The lowest score is 11 and the highest score is 77. High total scores from the scale indicate positive motherhood self-assessment. The Cronbach Alpha reliability coefficient of the Semantic Difference Scale-Me as a Mother scale was determined as 0.73-0.74.

CONTACTS AND LOCATIONS:
Overall Officials: Songül Kekil, Principal Investigator — Muş Hasköy Family Health Center; Sibel Öztürk, Asst. Prof., Study Director — Ataturk University Faculty of Health Sciences Department of Midwifery
Locations (1):
- Muş Hasköy Family Health Center, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No